CLINICAL TRIAL: NCT00497133
Title: Alpha-Cell Sensitivity to GLP-1 in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry); The Danish Diabetes Association (Other)
Responsible Party: K. J. Hare, Gentofte University Hospital, University of Copenhagen.
Other Study IDs: H-KA-20070023
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: glucoseintolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for further analyzes and buffy coat
Oversight: Data Monitoring Committee: No

SUMMARY:
Glucagon-like peptide 1 is known to improve sensitivity of the pancreatic beta-cell. Further it inhibit secretion from the pancreatic alpha-cell by mechanisms not fully understand. With this study we wish to elucidate the potential of GLP-1 to increase the sensitivity of the alpha-cell.

Type 2 diabetic patients and control subjects receive infusions of GLP-1 in increasing doses or saline, alpha- and beta-cell responses are measured in blood-samples. During the study plasma-glucose levels are clamped at fasting levels.

With this study we hope to elucidate the pathophysiology behind defect glucose tolerance in type 2 diabetes mellitus and further more the potential of GLP-1 in treatment of type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Background: Glucagon-like peptide-1 (GLP-1) possesses insulinotropic and glucagonostatic properties, and, therefore, GLP-based antidiabetic therapies have been developed. Even though the insulinotropic potency of GLP-1 has been shown to be reduced in patients with type 2 diabetes mellitus (T2DM), a small dose of GLP-1 is capable of normalizing the beta-cell responsiveness to glucose in these patients. The glucagonostatic potency of GLP-1 in patients with T2DM is not known, and, furthermore, the capability of GLP-1 to reestablish normal glucagon secretion in these patients remains to be elucidated.

Objective: To investigate the alpha-cell sensitivity to GLP-1 in patients with T2DM and to establish if GLP-1 is able to reestablish normal glucagon secretion in such patients.

Method: Ten patients with T2DM and ten healthy control subjects are clamped at their fasting blood glucose levels during GLP-1 infusions at increasing doses (0.25, 0.5, 1.0 and 2.0 pmol/kg/min) and placebo, respectively. Furthermore, the patients will be hospitalized overnight while receiving intravenous insulin and thereafter examined under normoglycaemic conditions. Blood are being drawn for analysis of plasma insulin, C-peptide, GLP-1 and glucagon.

Expected results and conclusions: We expect that GLP-1 will inhibit glucagon secretion in a dose dependent manner, leading too an increase in glucose turn-over. The results will potentially elucidate the interaction between GLP-1 and glucagon secretion and thereby broaden our knowledge on the pathophysiology of T2DM. Furthermore, the present study will determine the therapeutic impact of GLP-1 on the alpha-cell deficiency characterizing patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Caucasians aged > 18 years diagnosed with T2DM due to WHO criteria.
* Normal haemoglobin
* HbA1c 6-10%
* BMI 23-35 kg/m2

Exclusion Criteria:

* Hepatic disease, ALAT > 2 x normal.
* Diabetic nephropathy, (S-creatinine >130μM or albuminuria).
* Diabetic neuropathy (reported)
* Proliferative diabetic retinopathy (reported)
* Medical treatment that cannot be paused for 12 hours
* Insulin- or glitazon treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus and matched control subjects.
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Juul Holst, Professor, MD,MMSc, Study Director — University of Copenhagen, Department of Biomedical Sciences
Locations (1):
- Gentofte Hostital, Dep. og Internal Medicin F, Gentofte Municipality, Hellerup, Denmark